CLINICAL TRIAL: NCT04410120
Title: Impact of Asthma Exacerbations: A Qualitative Study
Brief Title: Impact of Asthma Exacerbations
Acronym: IMPAX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 20038
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Asthma Attack
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma with recent (<4/52) asthma attack
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Semi-structured 45 minute interviews regarding impact of asthma attacks

SUMMARY:
The purpose of the study is to gain a deeper understanding of the impact of asthma attacks on the lives of patients who experience them. This will help us to describe the true extent of the impact of asthma attacks on factors of importance to patients which have not previously been well described, including the psychological, social, financial and emotional burden of asthma attacks.

Additionally, it is hoped that detailed questioning regarding features of asthma attacks from a patient perspective will improve our understanding of patient recognition of attacks, consistency of certain features of attacks and patient views regarding preventative strategies for attacks. Patient experiences of asthma attacks are poorly described in previous research. Hence this work is expected to provide useful insights into these experiences which will contribute to improvements in detecting, treating and preventing asthma attacks.

The study will consist of a one-off interview lasting about 45 minutes with patients who have recently had asthma attacks. We plan to recruit patients for the study from an outpatient clinic for those who have had a recent attack or from a register of patients who have volunteered for future asthma research studies. The interviews will take place in person at the Respiratory Research Unit at the Nottingham City Hospital or over the telephone depending on patient preference.

ELIGIBILITY:
Inclusion Criteria:

* Adults with previous clinician diagnosis of asthma (16 years and above)
* Recent (≤4 weeks) asthma attack for which patient received ≥3 days of systemic corticosteroid treatment

Exclusion Criteria:

* Anyone under the age of 16 years.
* Anyone unable to speak or understand English.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with previous clinician diagnosis of asthma who have had a recent (≤4 weeks) asthma attack for which they received ≥3 days of systemic corticosteroid treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Thematic analysis of interview transcripts using framework approach | One off 45 minute interview
  Thematic analysis of interview transcripts using framework approach

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Respiratory Research Unit, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pradhan A, Jayes L, Bains M, Martin MJ. Patient experience, understanding and self-management of asthma attacks: a qualitative study. J Asthma. 2025 May;62(5):872-880. doi: 10.1080/02770903.2024.2449230. Epub 2025 Jan 10. PMID 39773014